CLINICAL TRIAL: NCT01909661
Title: Tolerancia a 2 fórmulas de Leche Infantil Altamente Hidrolizadas en Base a proteínas de Arroz y a caseína en niños Con Alergia a Las proteínas de Leche de Vaca
Brief Title: Tolerance of Infants With Cow's Milk Protein Allergy to Extensively Hydrolyzed Rice Protein or Casein Infant Formulas
Acronym: JUNGLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lactalis (Industry)
Collaborators: Biosearch S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LRD - 2013 - JUNGLO
Record Dates: First submitted 2013-07-18; First posted 2013-07-26 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2013-07

CONDITIONS: Cow Milk Protein Sensitivity; Tolerance; Growth Failure
Keywords: allergy; Cow's milk protein; Tolerance; Efficacy; Infants' growth
MeSH Terms: conditions — Failure to Thrive; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Damira/Celia peptide hydrolyzed casein (Experimental): Extensively Hydrolyzed (EH)casein infant formula
  Interventions: Other: Damira/Celia peptide hydrolyzed casein
- Picot riz/Celia rice/Sanutri arroz (Experimental): Picot riz/Celia rice/Sanutri arroz Extensively Hydrolyzed (EH) rice protein infant formula
  Interventions: Other: Picot riz/Celia rice/Sanutri arroz

INTERVENTIONS:
Other: Damira/Celia peptide hydrolyzed casein
  Arms: Damira/Celia peptide hydrolyzed casein
Other: Picot riz/Celia rice/Sanutri arroz
  Arms: Picot riz/Celia rice/Sanutri arroz

SUMMARY:
The objective of this double blinded randomized study is to assess the tolerance of two extensively protein hydrolyzed infant formulas, one based on rice protein and the other one on casein, at introduction, and after 3 months of consumption, and their efficacy on growth and on the reduction of allergy symptoms through a 3 months consumption period.

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy newborns (37-42 Weeks gestation)
* Weight at birth ≥ 2500 g
* Aged between birth to 9 months
* Symptoms of allergy (Skin or digetive)
* Suspicion of cow milk protein allergy
* Infants whose parents/caregivers/legal guardians have the ability to understand and comply with the requirements of the study
* Infants whose parents/caregivers/legal guardians gave their written informed consent to the infant's participation in the study

Exclusion Criteria:

* Children who have returned to breastfeeding
* Presence of any condition, that, in the opinion of the investigator is a contra-indication to the particpation of the infant in the study
* In the past 15 days, treatment or medication likely to :

  * induce confusion in the allergy tets (ex. : Skin Prick Test) and / or
  * mask the symptoms of an allergic reaction (Anti-allergy medications ; anti-histaminic, anti-leucotrienes, corticosteroids, …)
* Newbonrs presenting a chronic or a genetic malformation, or a chromosomal or other disease, that in the opinion of the investigator could mask the study results
* Children who show signs of malnutrition, or prolonged diarrhea
* Children whose parents show no willingness to comply with study requirements
* Consumption of soya protein based, hydrolyzed protein or elemental (amino acid) formula for more than 21 days before inclusion, unless the skin prick test to cow's milk protein is positive, and the IgE level indicates the existence of IgE mediated allergy to cow's milk protein.

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 114 (Actual)
Dates: Start 2013-03; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Proportion of infants who tolerate either the rice hydrolyzed protein infant formula or a hydrolyzed casein infant formula after 24h consumption. | 24h
  Tolerance is absence of clinical signs.

SECONDARY OUTCOMES:
Effectivness of the hydrolyzed protein formulas in terms of growth and allergy symptoms improvement. | 3 months
  Evaluate during 3 months of consumption the effectiveness of the formulas, in terms of :
  * infant growth, through anthropometric measures (body weight, length and head circumference)
  * allergy symptoms, through the improvement of the allergy symptoms.

OTHER OUTCOMES:
Volume of infant formula consumed by the infants | 3 months
  Volume of infant formula consumed by the infants in 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Biosearch S.A., Granada, Spain